# STATISTICAL ANALYSIS PLAN

# **BASICC**

# - PMCF study -

**Protocol:** LPH-2202

**Sponsor:** LALLEMAND PHARMA AG

Via Selva 2, 6900 Massagno, Switzerland

**CRO** in charge of the

**PHARMNDEV** 

**Monitoring:** 

Quai du Seujet 28 1201 Geneva, Switzerland

CRO in charge of the

**AXIODIS CRO** 

**Data-Management:** 

58 boulevard d'Arcole

31000 TOULOUSE, FRANCE

CRO in charge of the

AXIODIS CRO

**Statistical Analysis:** 

58 boulevard d'Arcole

31000 TOULOUSE, FRANCE

**Author:** Kévin CHAPDELAINE

**Version:** Final, Version 1.0

**Date:** August 09<sup>th</sup>, 2023

#### **CONFIDENTIAL MEDICAL DATA**

This document is the property of LALLEMAND PHARMA AG.

This document should not be amended, used or communicated without the prior written permission of LALLEMAND PHARMA AG.

# **HISTORY OF VERSIONS**

| Version<br>number | Date | Author | | Changes compared to the previous version |
|---|---|---|---|---|
| 01 | 09/08/2023 | K.<br>CHAPDELAINE | С | |

A: Addition, C: Creation, D: Deletion, M: Modification

AXIODIS CRO 2/47

# APPROVAL OF THE STATISTICAL ANALYSIS PLAN

| Protocol | LPH-2202 |
|----------|----------|

Meeting of the Committee of Validation

for the Data-Review

September 2023

Statistical Analysis Plan 09/08/2023

| D 9.994 | G: 4 | D 4 |
|-----------------------------|-----------|------|
| Responsibilities | Signature | Date |
| Kévin CHAPDELAINE | | |
| AXIODIS CRO | | |
| (Statistician) | | |
| kchapdelaine@axiodis.com | | |
| Catherine GENTIL | | |
| AXIODIS CRO | | |
| (Statistician reviewer) | | |
| cgentil@axiodis.com | | |
| Dr Frédéric DURMONT | | |
| (Sponsor's representative) | | |
| fdurmont@lallemand.com | | |
| Dr Rada MARKOVA | | |
| (Coordinating investigator) | | |
| rada_markova@yahoo.com | | |
| Sylvanie BONNET | | |
| (Clinical Study Lead) | | |
| sbonnet@pharmndev.ch | | |
| Géraldine JULOU-SCHAEFFER | | |
| (Clinical Project Manager) | | |
| gschaeffer@pharmndev.ch | | |

**AXIODIS CRO** 3/47

# LIST OF ABBREVIATIONS

AE: Adverse Event

ANCOVA: Analysis of covariance

ARSSQ: Acute Rhinitis Symptoms Severity Questionnaire
ATC: Anatomical Therapeutic Chemical Classification

AUC: Area Under the Curve
CI: Confidence Interval
CRF: Case Report Form

CRO: Contract Research Organisation

Dx: Day x

[E]: Number of eventsFAS: Full Analysis Set

ICH: International Conference on Harmonisation

LOCF: Last Observation Carried Forward

MedDRA: Medical Dictionary for Regulatory Activities
NSAID: Non-Steroidal Anti-Inflammatory Drugs

PMCF: Post-Market Clinical Follow-up

PP: Per Protocol
PT: Preferred Term

Q1 / Q3: First / Third Quartile

QoL: Quality-of-Life

SAS®: Statistical Analysis System

SD: Standard deviation SOC: System Organ Class

TEAE: Treatment-Emergent Adverse Event

Vy: Visit y

WHO-DRUG: World Health Organization Drug Dictionary

AXIODIS CRO 4/47

# **TABLE OF CONTENTS**

| 1. Introduction | |
|---|---|
| 2. Study objectives | 7 |
| 2.1. Primary objective | 7 |
| 2.2. Secondary objectives | 7 |
| 3. Study design | 7 |
| 4. Sample size | |
| 5. Definition of the analysis sets | 9 |
| 6. Statistical methods | |
| 6.1. Data processing | |
| 6.2. Description | |
| 6.3. Statistical/Analytical issues | |
| 6.3.1. Significance level | |
| 6.3.2. Interim analysis | |
| 6.3.3. Multiplicity | |
| 6.3.4. Multicentre studies and Adjustment for covariates | |
| 6.3.5. Handling of dropouts and missing data | |
| 6.4. General conventions and/or calculated variables | |
| 6.4.1. Patient reference start/end dates | |
| 6.4.2. Computation of a duration | |
| 6.4.3. Missing dates of inclusion visit or end of study | |
| 6.4.4. Missing start/end dates of adverse events / incidents | |
| 6.4.5. Missing start/end dates of concomitant medications | |
| 6.4.6. Scores of ARSSQ | 13 |
| 6.4.7. AUC on global score of ARSSQ | |
| 7. Study patients | |
| 7.1. Disposition of patients | |
| 7.2. Protocol deviations | |
| 7.3. Data Sets Analysed | |
| 8. Demographic and other baseline characteristics | |
| 8.1. Demographic characteristics | |
| 8.2. Previous medications | |
| 8.3. Medical and surgical past history | |
| 8.4. Acute Rhinitis Symptoms Severity Questionnaire | |
| 8.5. Other baseline variables | |
| 9. Compliance | |
| 10. Efficacy | |
| 10.1. Analysis of the primary efficacy criterion | |
| 10.2. Analysis of the secondary efficacy criteria | |
| 10.2.1. Modelling of AUC on global score by multivariate ANCOVA | |
| 10.2.2. Durations of cold symptoms and of impacts on Quality-of-Life | |
| 10.2.3. Use and number of days of use of conventional common cold medications | |
| 10.3. Concomitant treatments | |
| 10.4. Non-related adverse events | |
| 11. Safety | |
| 11.1. Treatment and study duration | |
| 11.2. Incidents | 24 |

| 12. Char | ges in the conduct of the study or planned analysis | 25 |
|---|---|---|
| | endices | |
| | List of statistical tables, figures and listings | |
| | Mock tables | |
| 13.3. | Acute Rhinitis Symptoms Severity Questionnaire – Daily report | 47 |

AXIODIS CRO 6/47

# 1. Introduction

This statistical analysis plan is based on protocol LPH-2202 – version 1.1, dated on February 2<sup>nd</sup>, 2023. It defines populations of analysis and the evaluation methods of the principal and secondary criteria.

Study Number: LPH-2202

**BASICC** 

# 2. STUDY OBJECTIVES

# 2.1. Primary objective

The primary objective is to assess the efficacy of **Healsea® Babykids** on the overall health status score of the Acute Rhinitis Symptoms Severity Questionnaire (ARSSQ) in 2-6 years old children during a treatment period of 7 to 10 days as compared to Placebo.

# 2.2. Secondary objectives

The secondary objectives are:

- To assess the impact of **Healsea® Babykids** on the duration of each infectious rhinitis symptom and on quality of life as compared to Placebo;
- To assess the impact of **Healsea**<sup>®</sup> **Babykids** on the intake of conventional common cold medications (antibiotics, antipyretics, mucolytics, decongestants, antitussives, systemic and topical corticosteroids) as compared to Placebo;
- Safety: to assess systemic and local tolerance of **Healsea**® **Babykids** over the study period.

#### 3. STUDY DESIGN

This is a prospective, interventional, double-blinded, placebo controlled, randomized, national (Bulgaria), multicentre PMCF study.

The study comprises two parts:

- Part 1 (D1-D11): treatment of the acute phase, with **Healsea**® **Babykids** or with **isotonic nasal spray** (**Placebo**), 2 puffs in each nostril 2 times per day with a minimum of 7-day-treatment period (14 intakes of the investigational device) up to 10 days (20 intakes of the investigational device);
- Part 2 (up to D15/D18): follow-up phase.

Investigational plan description (see Figure 1):

# - Visit 1 (V1) – (Day 1): Screening/Inclusion/Randomization

Information and provision of the information sheet to legal guardians/parents of participants, consent signature, demographic data and medical history, ongoing medication, inclusion/non-inclusion criteria, physical and clinical examination, baseline assessment of the ARSSQ, randomization, diary presentation, treatment dispensation of **Healsea**® **Babykids** Nasal Spray or **Placebo (Isotonic nasal spray)** (according to randomization list).

AXIODIS CRO 7/47

#### **D1-D8 up to D1-D11 (at home):**

Daily completion of the paper diary (questionnaire, adverse events/incidents and concomitant medications), Healsea® Babykids / Placebo nasal spray treatment daily administration.

# Between D8 and D11 (at home):

End of Healsea® Babykids / Placebo nasal spray treatment.

# Up to D15/D18 (at home):

Daily completion of the diary (adverse events/incidents, concomitant medications, ARSSQ if applicable, until the patient feels not sick for two consecutive days).

#### Visit 2(V2) - (Day 15-18): end of study

Diary review, reporting of the adverse events/incidents, compliance, ARSSQ completion if "not sick" is not ticked for two consecutive days in the previous days.

The maximal study duration for each patient is 18 days.

| | Acute p | Acute phase Follow-up phase | | phase |
|---|---|---|---|---|
| Visit name | Screening/Inclusion | At home | At home | End of study |
| Visit Number | V1 | | *************************************** | V2 |
| Days | D1 | D1 to D11 | D12 to End of study | D15-D18 |
| Informed consent | х | | | |
| Eligibility criteria | х | | | |
| Demography and Medical history *** | x | | | |
| Physical and clinical examination | x | | | x |
| Baseline assessment of the Acute Rhinitis Symptoms<br>Severity Questionnaire | х | | | |
| Ongoing medication | x | | | |
| Randomization | х | | | |
| Treatment (Healsea® Babykids or Placebo) | Х* | Χ# | | |
| Subject paper diary (Acute Rhinitis Symptoms Severity<br>Questionnaire**) | | | | |
| Adverse events/incidents and concomitant medication reporting | | | | |
| Compliance | | | | x |

Figure 1: Flow chart of the study

**AXIODIS CRO** 8/47

<sup>\*</sup> Treatment dispensation

\*\* ARSSQ to be completed with the investigator on site at screening and at the end of the study if the patient still has symptoms ("not sick" not ticked for 2 consecutive days in the previous days). After day 8, until complete resolution of symptoms for 2 consecutive days (question 1 of the questionnaire).

<sup>#</sup> Treatment from D1 to D8 and up to D11.
\*\*\* Medical History - Relevant medical history in connection to infectious acute rhinitis, allergic rhinitis, nasal disorders and asthma back to 2 years

### 4. SAMPLE SIZE

This is a PMCF study. The primary endpoint is a customized symptom and quality of life questionnaire. An arbitrary cohort of 200 children has been chosen. A cohort of 100 children in the Healsea® Babykids arm and 100 children in the Placebo arm is anticipated to allow to demonstrate the interest of using Healsea® Babykids in the acute infectious rhinitis. Indeed, 100 patients by arm are enough to detect a Cohen's effect size of 0.4 with a power of 80% and a type I error of 5%. Cohen's effect size is defined as the standardized difference between area under the curve (AUC) in groups. According to Cohen's methodology, 0.4 is an intermediate size between a small effect (0.2) and a medium effect (0.5) and is coherent with the expected result. The Placebo arm will be used as the reference group.

Study Number: LPH-2202

BASICC

The recruitment will be performed using a 1:1 randomization ratio.

# 5. DEFINITION OF THE ANALYSIS SETS

Enrolled patients: all patients whose parents/legal guardians signed an informed consent.

Included patients: all the enrolled patients who participated in the study.

Randomised patients: all the included patients who were assigned a treatment number.

Safety population: all the randomised patients who used the nasal spray at least once.

Full Analysis Set (FAS): all the patients from the Safety population and with at least one postbaseline efficacy data.

Any patient not satisfying major entry criteria or for whom post randomisation data are not available will be identified by the Validation Committee during the data review, and could be excluded from the FAS in agreement with circumstances exposed in the ICH-E9 §5.2.1.

Per Protocol (PP) Set: Efficacy population based on the FAS without patients with major protocol deviations.

The status of protocol deviations (minor or major) will be validated during the data review meeting.

Safety endpoint will be performed on the Safety Set.

The analyses of primary and secondary endpoints will be performed on the FAS.

The primary and one secondary (modelling of AUC on global ARSSQ score by multivariate ANCOVA) endpoints will also be analysed on the PP set, analyses on the PP set being supportive in superiority trials.

**AXIODIS CRO** 9/47

# 6. STATISTICAL METHODS

#### 6.1. Data processing

The analyses will be computed with SAS Version 9.4 TS Level 1M6 Copyright (c) 2016 by SAS Institute Inc., Cary, NC, USA.

# 6.2. Description

The number of available data and the number of missing data will be given and the following descriptive statistics will be provided:

- For <u>quantitative parameters</u>: mean, standard deviation, median, Q1, Q3, extreme values (min and max).
  - In this case, calculated statistics (mean, standard deviation, median, Q1, Q3) will generally be displayed with one more significant figure than the observed data, unless the described variable necessitates less precision.
- For <u>qualitative parameters</u>: number and percentage of each modality.
   Usually, one decimal digit will be given. A second decimal digit could be provided to improve the display, if required.

#### 6.3. Statistical/Analytical issues

#### 6.3.1. Significance level

All statistical analyses will be performed at the 0.05 global significance level (type I error rate), using two-sided tests.

The statistical results will only allow to conclude on the primary efficacy criterion. All other statistical results have to be considered within a descriptive perspective and not as inferential issues. No adjustment for Type I error will be done. P-values of statistical tests on secondary criteria will be provided for information only.

#### 6.3.2. Interim analysis

No interim analysis will be performed.

#### 6.3.3. Multiplicity

There is only one main efficacy criterion and no comparative testing will be performed, then multiplicity adjustments are not needed.

# 6.3.4. Multicentre studies and Adjustment for covariates

No adjustment on centre will be performed.

AXIODIS CRO 10/47

# 6.3.5. Handling of dropouts and missing data

# a) Repositioning of visits

Not applicable.

# b) Partially filled scales and missing data (other than ARSSQ and dates)

Concerning dates and ARSSQ, see §6.4.

No imputation will be done. Missing data will not be estimated and will be treated as missing data for the statistical analysis.

# c) Dropouts

Patients from FAS who prematurely discontinued the study will be included in the analysis.

Except for ARSSQ and dates, no method will be applied to replace missing data.

# 6.4. General conventions and/or calculated variables

# 6.4.1. Patient reference start/end dates

For each patient, the reference dates will be the following:

- The <u>reference start date</u> is the date of inclusion visit.
- The <u>reference end date</u> is the date when patient was determined to have ended the trial.

# 6.4.2. Computation of a duration

The formula below will be generally used:

- Duration (in days) = Date#2 - Date#1 + 1 day

# 6.4.3. Missing dates of inclusion visit or end of study

Missing dates of inclusion visit and of end of study will be reviewed by the members of the Validation Committee and extrapolated using all information recorded.

AXIODIS CRO 11/47

# 6.4.4. Missing start/end dates of adverse events / incidents

In the following paragraphs, adverse events and incidents will be referred to as "adverse events" for ease of reading.

# a) Start date

Completely missing date: it will be estimated by the reference start date.

#### If the day and the month are missing:

- If the year = year of reference start date, it will be estimated by the reference start date
- If the year < year of reference start date, it will be estimated by the 31st December
- If the year > year of reference start date, it will be estimated by the 1st January

# If only the day is missing:

- If the month/year = month/year of reference start date, it will be estimated by the date of reference start date
- If the month/year < month/year of reference start date, it will be estimated by the last day of the month
- If the month/year > month/year of reference start date, it will be estimated by the first day of the month

If after imputation, the estimated start date is after the end date of the adverse event, it will be replaced by the end date of the adverse event.

# b) End date

Note: the following rules concern events that are not "ongoing" at the end of the study.

Completely missing date: it will be estimated by the reference end date

### If the day and the month are missing:

- If the year = year of reference end date, it will be estimated by the reference end date
- If the year < year of reference end date, it will be estimated by the 31st December
- If the year > year of reference end date, it will be estimated by the 1<sup>st</sup> January

# If only the day is missing:

- If the month/year = month/year of reference end date, it will be estimated by the reference end date
- If the month/year < month/year of reference end date, it will be estimated by the last day of the month
- If the month/year > month/year of reference end date, it will be estimated by the first day of the month

If after imputation, the estimated end date is before the start date of the adverse event, it will be replaced by the start date of the adverse event.

AXIODIS CRO 12/47

# 6.4.5. Missing start/end dates of concomitant medications

Same rules as for adverse events.

#### 6.4.6. Scores of ARSSQ

To compute any score of ARSSQ, if the questionnaire has been completed at a given time point except some items, these missing answers will be imputed by the last observation carried forward (LOCF).

At time points the questionnaire has not been completed at all, no imputation will be done and the score will be missing.

# 6.4.7. AUC on global score of ARSSQ

The computation of the AUC on global score of the questionnaire will be made for patients with non-missing value at D1 and at least another non-missing time point between D2 and D11. Otherwise, the AUC will be missing.

The AUC will be computed by the trapezoidal rule from D1 to D11 (Acute Phase).

If the value at D11 is missing, then it will be estimated by the value at the last non-missing time point before D11.

AXIODIS CRO 13/47

### 7. STUDY PATIENTS

#### 7.1. Disposition of patients

Enrolled patients as well as included and randomised patients will be summarised using frequencies and percentages.

The number and percentage of patients who withdrew prematurely after inclusion, are lost to follow-up as well as the number of completers will be described by treatment group and overall. All withdrawn patients after their inclusion will be described regarding their main reason for withdrawal.

#### 7.2. Protocol deviations

Protocol deviations will be discussed during the data review meeting and the status (minor or major) of these deviations will be validated in order to identify the patients to be excluded from the Per Protocol Set.

Major deviations are defined by:

- Non-compliance with the inclusion or exclusion criteria;
- No assessment of the primary efficacy criterion (ARSSQ) at D1, D5±1 and D8-1 during the treatment period;
- Intake of forbidden medication: saline irrigation;
- Intake of wrong treatment, i.e. wrong treatment given to the patient after randomization;
- A compliance to study product intake below 80% or greater than 120%;
- More than 23 intakes of Babykids nasal spray.

All other deviations will a priori be considered as minor, e.g.:

- V2's date that does not conform with the flow chart of the study;
- V2 not performed;
- Treatment stopped before D8 morning or after D11 morning (less than 14 intakes of the investigational device or more than 20 intakes);
- ARSSQ data missing (but data available at D1, D5±1 and D8-1) until patient's recovery (two consecutive and negative "not sick" answers to the first item) or D18/patient's end of study, whichever occurs first.

Major and minor deviations and their types will be described by treatment group and overall. They will be summarised with frequencies and percentages.

Patients will be counted only once within each type of deviation and within each category (major/minor).

A listing of all deviations will be provided for all included patients, including the category.

# 7.3. Data Sets Analysed

The number and percentage of patients in each analysis data set, as described in §5, will be provided.

AXIODIS CRO 14/47

Statistical Analysis Plan

### 8. Demographic and other baseline characteristics

All demographic and baseline characteristics will be described on the Safety Set and on the FAS, by treatment group and overall.

**BASICC** 

# 8.1. Demographic characteristics

Age (years) and sex will be summarised using descriptive statistics already mentioned in §6.2. Age will be computed using the formula below:

Age (years) = Collected Age (years) + [Age precision in months] / 12 (rounded at 1 digit)

#### 8.2. Previous medications

Previous and concomitant medications (taken at least once before reference start date) are coded by ATC class and substance name using the WHO-DRUG dictionary version 2022 Q1.

They will be summarised with frequencies and percentages.

Patients will be counted only once within these ATC categories.

Moreover, answers to questions about past or concomitant forbidden medications and about concomitant treatments for first symptoms of infectious rhinitis will be summarised.

# 8.3. Medical and surgical past history

Medical and surgical past history is coded using the MedDRA dictionary version 25.0. Events are classified by System Organ Class and Preferred Term.

The number and percentage of patients with at least one medical and surgical past history of each category (SOC/PT) will be given.

Patients will be counted only once within these categories.

#### 8.4. Acute Rhinitis Symptoms Severity Questionnaire

The scores to each of the ten items of the ARSSQ, the score of cold symptoms (the sum of the scores to the items 2 to 7), the score of impact on Quality-of-Life (the sum of the scores to the items 8 to 10) and the global score (the sum of the scores to all the ten items) will be described at baseline.

A Student (or Wilcoxon if the normality assumption is not acceptable) between-groups test will be performed for each score.

#### 8.5. Other baseline variables

The presence of fever in the patient and the reported body temperature will be summarised. The presence of fever in each group will be compared by means of chi-square or exact Fisher test.

A Student (or Wilcoxon if the normality assumption is not acceptable) between-groups test will be performed for the reported body temperature.

AXIODIS CRO 15/47

# 9. COMPLIANCE

Compliance will be calculated according to the following formula and analysed on the Safety set, by treatment group and overall.

The compliance will be calculated as follows:

Compliance (%) = [Initial weight of the container (g) – Real weight of the container at the end of the study (g)]  $\times$  100 / [Initial weight of the container (g) – Theoretical weight of the container at the end of complete study (g)]

with:

- Initial weight of the container = 32.615 g;
- Theoretical weight of the container at the end of complete study is a function of treatment duration and is noted *weight*<sub>theo</sub>;

i.e.:

Compliance (%) = 
$$100 \times \frac{32.615 - weight_{end}}{32.615 - weight_{theo}}$$

with weightend the real weight of the container at the end of the study in g.

The table below gives the value of  $weight_{theo}$  by last day of treatment:

Table 1: Theoretical weight of the container at the end of complete study by last day of treatment

| Patient stopped treatment | weighttheo (g) |
|---------------------------|----------------|
| Before D8 | 27.55875 |
| At D8 morning | 27.55875 |
| At D8 evening | 27.21750 |
| At D9 morning | 26.85750 |
| At D9 evening | 26.53750 |
| At D10 morning | 26.21500 |
| At D10 evening | 25.87125 |
| At D11 morning | 25.52500 |
| At D11 evening | 25.20250 |
| At D12 morning | 24.86500 |
| At D12 evening | 24.51000 |
| After D12 | 24.51000 |

Compliance will be also described according to the following categories: <80%, [80%; 120%] and >120%.

Note that in case of spray not returned, compliance will be considered unknown and missing.

AXIODIS CRO 16/47

# 10. EFFICACY

# 10.1. Analysis of the primary efficacy criterion

The primary objective will be analysed by performing a t-test (or a Wilcoxon test if the normality assumption is not acceptable) on the means of AUC on global score of ARSSQ during the first eleven days of the study between treatment groups.

The answers of the ten items of ARSSQ are scored <u>from 0 to 3</u> (0: negative answer; from 1 to 3: positive answer with an increasing severity level). See the daily report in appendix (§13.3). The global ARSSQ score at each time point is the sum of the scores to the ten items of the ARSSQ:

At each time point t: ARSSQTOT(t) = 
$$\sum_{j \text{ in } \{1; ...; 10\}} ARSSQ_j(t)$$

AUC of global ARSSQ score will be computed by the method described in §6.4.7.

Patients will be analysed on the FAS and the PP Set. In each case, boxplots of the AUC on global score will be realized by treatment group. The number of available data and the p-value will be printed on the figure.

#### 10.2. Analysis of the secondary efficacy criteria

The analysis of the secondary efficacy criteria will involve multivariate analysis.

The selection of variables in multivariate analysis will be performed using a 0.20 significance level and a stepwise method. Covariates considered as potential confounding factors to be initially tested with the treatment in the multivariate models are:

- Body temperature at baseline (°C);
- Scores to each of the items 2 to 7 of the ARSSO at baseline.

All multivariate analyses below will follow this logic.

# 10.2.1. <u>Modelling of AUC on global score by multivariate ANCOVA</u>

A multivariate ANCOVA model of the AUC on global score of ARSSQ during the first eleven days of the study will be performed.

Patients will be analysed on the FAS and the PP Set.

AXIODIS CRO 17/47

# 10.2.2. Durations of cold symptoms and of impacts on Quality-of-Life

Hereinafter, the "recovery date" is the first day of the <u>two</u> first <u>consecutive</u> days the patient gave a negative answer to the question 1 ("not sick") without giving a positive answer to the same question (other than "not sick") later. Otherwise, there is no "recovery date" for the patient.

The scores of cold symptoms and of impact on Quality-of-Life (QoL) will be computed at each time-point the patient completed the questionnaire (see §6.4.6), using the following formulae:

At each time point t: ARSSQ<sub>SYMP</sub>(t) = 
$$\sum_{j \text{ in } \{2; ...; 7\}} ARSSQ_{j}(t)$$
  
ARSSQ<sub>QOL</sub>(t) =  $\sum_{j \text{ in } \{8; ...; 10\}} ARSSQ_{j}(t)$ 

• The <u>duration of common cold</u> is defined as the duration between the reference start date and the recovery date.

# Common cold's duration (days) = Recovery date – Reference start date

The origin date will be the reference start date.

The considered event is the end of common cold, i.e. the recovery of the patient. The event date will be the last day before the recovery date.

Patients without recovery date will be censored at D18 or at the end of the study, and the censoring date will be the date of D18 or the reference end date, whichever occurs first.

• The <u>duration of the cold symptoms</u> is defined as the duration between first symptomatic day and last symptomatic day.

#### Cold symptom's duration (days) = Last symptomatic day - first symptomatic day + 1

The first symptomatic day is the first day the patient had a non-zero and non-missing score of cold symptoms. It will be the origin date.

The last symptomatic day is defined as the day before the <u>two</u> first <u>consecutive</u> days the patient had a zero score of cold symptoms without having a non-zero and non-missing score of cold symptoms later. The considered event is the end of cold

AXIODIS CRO 18/47

symptoms, i.e. the definitive nullification of the corresponding score during at least two consecutive days.

The considered symptomatic days are between D1 and either D18, or the end of the study, or the day before the recovery date, whichever occurs first. Symptomatic days from the recovery date will not be taken into account.

For patients who definitely nullified the score of cold symptoms, or for patients with a recovery date, the event date will be the last day before the definitive nullification of the score of cold symptoms, or before the recovery date if it exists.

Patients who did not definitely nullify the score of cold symptoms, and without recovery date, will be censored at D18 or at the end of the study, and the censoring date will be the date of D18 or the reference end date, whichever occurs first.

For patients who never had a non-zero score of cold symptoms (never ticked "mild", "moderate" or "severe" for any symptom) and having completed the questionnaire at D1, the origin date for the symptom will be D1, the cold symptoms will be censored at D1 and the duration will be zero. If patients who never reported the presence of any symptom did not complete the questionnaire at D1, neither origin date nor censoring date will be defined for cold symptoms and the duration will be missing.

• The <u>duration of impact on QoL</u> is defined as the duration between first impacted day and last impacted day.

# Impact on QoL's duration (days) = Last impacted day – first impacted day + 1

The first impacted day is the first day the patient had a non-zero and non-missing score of impact on QoL. It will be the origin date.

The considered event is the end of impact on QoL, i.e. the definitive nullification of the corresponding score during at least two consecutive days. The last impacted day is defined as the day before this definitive nullification, and the duration is computed by the same way as for cold symptoms' duration.

A Cox survival regression model will be used to analyse each of the durations of common cold, of cold symptoms and of impact on QoL.

Since the computed duration in the three cases is a recovery time and not a survival time, unlike the usual case of application of Cox survival regression, the provided hazard ratios will measure the likeliness of the recovery.

Consequently, and particularly for the treatment (with Placebo as reference), a hazard ratio greater than 1 will have to be considered under a positive aspect, because it will significate that the recovery is more likely under Healsea<sup>®</sup> Babykids treatment than under Placebo. On the contrary, a hazard ratio lower than 1 will have to be considered under a negative aspect.

For the three durations, a forest plot of the hazard ratios and their 95% CIs from the final multivariate Cox survival regression model will be provided.

AXIODIS CRO 19/47

In addition, for the three durations, a Kaplan-Meier graph will be provided. Survival curves will be drawn by treatment group. Number of sick / symptomatic / impacted patients, number of events (recoveries) and number of censors in each arm will be displayed on the same graph, as well as the log-rank p-value.

For the same reason as above and unlike the usual case of application of Kaplan-Meier graph, if the log-rank p-value is under 5%, a survival curve for Healsea<sup>®</sup> Babykids group under the curve for Placebo group will have to be considered under a positive aspect, and the contrary under a negative aspect.

Patients will be analysed on the FAS.

AXIODIS CRO 20/47

Statistical Analysis Plan

# 10.2.3. <u>Use and number of days of use of conventional common cold</u> medications

A multivariate logistic regression model will be used to analyse use (yes/no) of conventional common cold medications (overall and by therapeutic class: antibiotics, antipyretics, mucolytics, decongestants, antitussives, systemic and topical corticosteroids).

BASICC

A multivariate Poisson regression model will be used to analyse the number of days of use of conventional common cold medications (overall and by therapeutic class).

The number of days of use of these medications is defined as follows:

- A day is counted when the patient used at least one of these medications this day;
- Each day is counted once, whatever the number of these medications used this day;
- The total number is the sum of all distinct days of use of these medications, from D1 to D18.

Patients will be analysed on the FAS.

#### 10.3. Concomitant treatments

Concomitant treatments are coded using the WHO-DRUG dictionary version 2022 Q1.

All treatments taken at least once from reference start date or appeared during the study will be summarised by Anatomical Therapeutic Class (ATC) and substance name. The number and percentage of patients in each category will be computed.

Patients will be counted only once within these ATC categories. They will be analysed on the FAS, by treatment group and overall.

Note: A medication which began strictly before reference start date and is on-going after reference start date is counted only in "previous medications" (see §8.2) and not in "concomitant medications".

AXIODIS CRO 21/47

# 10.4. Non-related adverse events

In the following paragraph, for a smoother reading:

- adverse events will be referred as AE;
- treatment-emergent adverse events will be referred as TEAE.

Adverse events are coded using the MedDRA dictionary version 25.0. They are classified by System Organ Class and Preferred Term.

For efficacy analyses, only non-related AEs are considered, i.e. adverse events with a relationship to study device equal to "not related". These analyses will be performed on the Safety Set and on the FAS, by treatment group and overall.

An adverse event will be considered as a treatment-emergent adverse event (TEAE) if:

- it was reported at least one day after screening;
- it was not present prior to the reference start date;
- it was present prior to the reference start date and worsened during the study (increase of intensity);
- it reappears after the reference start date (finished before the reference start date).

Missing or incomplete dates will be estimated as described in §6.4.4 in order to determine the TEAEs, but they will be <u>presented as reported in CRF in the data listings</u>. Generally, an adverse event for which the onset date is missing or incomplete and does not permit to identify the onset according to the date of the reference start date (i.e. missing onset day and month/year corresponding to the reference start date) will be considered as treatment-emergent.

<u>Note</u>: if the intensity/severity is missing, a conservative approach will be adopted and the intensity/severity will be considered as severe.

A given treatment-emergent adverse event (according to the MedDRA terminology) will be counted only once per patient. If a patient experienced several AEs in the same SOC/PT, the most severe intensity will be retained for this SOC/PT.

#### Summary of non-related adverse events

A summary table will be produced:

- number and percentage of patients with at least one non-related adverse event (AE);
- number and percentage of patients with at least one non-related AE leading to definitive study device discontinuation;
- number and percentage of patients with at least one non-related AE leading to definitive study discontinuation;
- number and percentage of patients with at least one serious non-related AE;
- number and percentage of patients with at least one non-related TEAE;
- number and percentage of patients with at least one serious non-related TEAE.

The number of non-related AEs of each category will also be provided in this table.

AXIODIS CRO 22/47

Statistical Analysis Plan Final version – August 09th, 2023

# Analysis of non-related treatment-emergent adverse event

The number and percentage of patients with non-related TEAEs will be summarised by System Organ Class and Preferred term.

The number of non-related TEAEs of each category will also be provided in this table.

A listing of serious non-related AEs will be provided.

All non-related AEs leading to definitive discontinuation of the trial device or to definitive discontinuation of the study will be listed.

AXIODIS CRO 23/47

# 11. SAFETY

The following analyses will be performed on the Safety Set, by treatment group and overall.

# 11.1. Treatment and study duration

Study duration will be calculated according to the formula below:

#### Study duration (days) = Reference End Date – Reference Start Date + 1

Treatment duration will be calculated according to the formula below:

#### Treatment duration (days) = Device Stop Date - Reference Start Date + 1

Both will be described (see §6.2) on the Safety Set.

In addition, number and percentages of patients who stopped treatment before D8, at D8 morning, at D8 evening, ..., at D12 morning, at D12 evening and after D12 will be provided.

#### 11.2. Incidents

For safety analyses, only incidents are considered, i.e. adverse events with a relationship to study device other than "not related".

#### Summary of incidents

A summary table will be produced:

- number and percentage of patients with at least one incident;
- number and percentage of patients with at least one incident leading to definitive study device discontinuation;
- number and percentage of patients with at least one incident leading to definitive study discontinuation;
- number and percentage of patients with at least one serious incident.

The number of incidents of each category will also be provided in this table.

#### Analysis of incident

The number and percentage of patients with incidents will be summarised by System Organ Class (SOC) and Preferred term (PT).

The number of incidents of each category will also be provided in this table.

A listing of serious incidents will be provided.

All incidents leading to definitive discontinuation of the trial device or to definitive discontinuation of the study will be listed.

AXIODIS CRO 24/47

# 12. CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSIS

The planned analysis in the protocol to assess the primary objective (multivariate ANCOVA model of the AUC on global score of ARSSQ during the first eleven days of the study) has been replaced by the comparison of the means of the AUC on global score of ARSSQ during the first eleven days of the study between treatment groups. The multivariate ANCOVA has been put among secondary analyses.

This change has no impact on the relevance of the sample size calculation since the primary endpoint is the same as planned in the protocol.

Moreover, since several patients still reported having symptoms while they reported they did not feel sick anymore at the question 1 during at least the two last days of completion of the ARSSQ, their positive answers to the cold symptoms' items have been considered as non-significant. Consequently, the question 1 has been taken into account in addition to the corresponding items to determine the end of the cold symptoms' duration, however only on the condition that the last days of completion were consecutive.

If the last days of completion were not consecutive, positive answers to cold symptoms' items are still considered as symptomatic, even if the two last answers to the question 1 are negative. The symptom ends at the last symptomatic day if the patient reported the absence of this symptom at least twice and consecutively after this day. Otherwise, the duration of the symptom is censored at D18 or at the end of the study, whichever occurs first.

The same change has been applied to compute the duration of impact on QoL.

AXIODIS CRO 25/47

# 13. APPENDICES

# 13.1. List of statistical tables, figures and listings

Study Number: LPH-2202

**BASICC** 

| File (BASICC) | Type | Number | Title | Mock |
|---|---|---|---|---|
| STUDY PATIENTS | | | | |
| T_14_1_1_1_ds_enrl.rtf | Table | 14.1.1.1 | Patients' disposition – Enrolled patients | T1 |
| F_14_1_1_ds_enrl.rtf | Figure | 14.1.1.1 | Patients' disposition – Enrolled patients | F1 |
| T_14_1_1_2_1_dv_incl.rtf | Table | 14.1.1.2.1 | Summary of protocol deviations by category and type – Included patients | T2 |
| L_14_1_1_2_1_dv_incl.rtf | Listing | 14.1.1.2.1 | Patients with at least one protocol deviation – Included patients | L1 |
| T_14_1_1_2_2_disc_incl.rtf | Table | 14.1.1.2.2 | Premature withdrawal – Reason of withdrawal | Т3 |
| L_14_1_1_2_2_disc_incl.rtf | Listing | 14.1.1.2.2 | Patients prematurely withdrawn – Included patients | L2 |
| DEMOGRAPHIC AND OTHER | BASELIN | E CHARACTER | ISTICS, COMPLIANCE, STUDY DURATION | |
| T_14_1_2_1_1_dm_saf.rtf | Table | 14.1.2.1.1 | Demographic characteristics – Safety Set | T4 |
| T_14_1_2_1_2_dm_fas.rtf | Table | 14.1.2.1.2 | Demographic characteristics – Full Analysis Set | T4 |
| T_14_1_2_2_1_1_prevm_saf.rtf | Table | 14.1.2.2.1.1 | Summary of previous medications – Safety Set | T5 |
| T_14_1_2_2_1_2_prevm_fas.rtf | Table | 14.1.2.2.1.2 | Summary of previous medications – Full Analysis Set | T5 |
| T_14_1_2_2_1_forbidm_saf.rtf | Table | 14.1.2.2.2.1 | Past or concomitant forbidden medications at baseline – Safety Set | Т6 |
| T_14_1_2_2_2_forbidm_fas.rtf | Table | 14.1.2.2.2.2 | Past or concomitant forbidden medications at baseline – Full Analysis Set | Т6 |
| T_14_1_2_2_3_1_cmbl_saf.rtf | Table | 14.1.2.2.3.1 | Concomitant treatments for first symptoms of infectious rhinitis at baseline – Safety Set | Т7 |
| T_14_1_2_2_3_2_cmbl_fas.rtf | Table | 14.1.2.2.3.2 | Concomitant treatments for first symptoms of infectious rhinitis at baseline – Full Analysis Set | Т7 |
| T_14_1_2_3_1_mh_saf.rtf | Table | 14.1.2.3.1 | Medical and surgical past history – Safety Set | Т8 |

AXIODIS CRO 26/47

Study Number: LPH-2202

BASICC

Statistical Analysis Plan
Final version – August 09th, 2023

| File (BASICC) | Туре | Number | Title | Mock |
|---|---|---|---|---|
| T 14 1 2 3 2 mh fas.rtf | Table | 14.1.2.3.2 | Medical and surgical past history – Full Analysis Set | Т8 |
| T 14 1 2 4 1 arssqbl saf.rtf | Table | 14.1.2.4.1 | Acute Rhinitis Symptoms Severity Questionnaire at baseline – Safety Set | Т9 |
| T 14 1 2 4 2 arssqbl fas.rtf | Table | 14.1.2.4.2 | Acute Rhinitis Symptoms Severity Questionnaire at baseline – Full Analysis Set | Т9 |
| T 14 1 2 5 1 fever saf.rtf | Table | 14.1.2.5.1 | Fever and body temperature at baseline – Safety Set | T10 |
| T_14_1_2_5_2_fever_fas.rtf | Table | 14.1.2.5.2 | Fever and body temperature at baseline – Full Analysis Set | T10 |
| T_14_1_3_compl_saf.rtf | Table | 14.1.3 | Summary of compliance per treatment group – Safety Set | T11 |
| T_14_1_4_stdur_saf.rtf | Table | 14.1.4 | Treatment and study durations by patient – Safety Set | T12 |
| EFFICACY | | _ | | |
| T 14 2 1 1 aucarssq_fas.rtf | Table | 14.2.1.1 | AUC on global score of ARSSQ per treatment group – Full Analysis Set | T13 |
| T_14_2_1_2_aucarssq_pp.rtf | Table | 14.2.1.2 | AUC on global score of ARSSQ per treatment group – Per Protocol Set | T13 |
| F_14_2_1_1_aucarssq_fas.rtf | Figure | 14.2.1.1 | Boxplots of AUC on global score of ARSSQ by treatment group – Full Analysis Set | F2 |
| F 14 2 1 2 aucarssq pp.rtf | Figure | 14.2.1.2 | Boxplots of AUC on global score of ARSSQ by treatment group – Per Protocol Set | F2 |
| T_14_2_2_1_1_ancovarssq_fas.rtf | Table | 14.2.2.1.1 | Multivariate ANCOVA model for the AUC on global score of ARSSQ – Full Analysis Set | T14 |
| T 14 2 2 1 2 ancovarssq pp.rtf | Table | 14.2.2.1.2 | Multivariate ANCOVA model for the AUC on global score of ARSSQ – Per Protocol Set | T14 |
| T_14_2_2_1_coxcc_fas.rtf | Table | 14.2.2.2.1 | Cox survival regression model for the duration of common cold – Full Analysis Set | T15 |
| F_14_2_2_2_1_1_hrcc_fas.rtf | Figure | 14.2.2.2.1.1 | Forest plot of Hazard Ratios from final multivariate Cox survival regression model for the duration of common cold – Full Analysis Set | F3 |
| F_14_2_2_2_1_2_kmcc_fas.rtf | Figure | 14.2.2.2.1.2 | Kaplan-Meier graph for the duration of common cold by treatment group – Full Analysis Set | F4 |
| T_14_2_2_2_coxcs_fas.rtf | Table | 14.2.2.2.2 | Cox survival regression model for the duration of cold symptoms – Full Analysis Set | T15 |

AXIODIS CRO 27/47

| File (BASICC) | Type | Number | Title | Mock |
|---|---|---|---|---|
| F_14_2_2_2_1_hrcs_fas.rtf | Figure | 14.2.2.2.1 | Forest plot of Hazard Ratios from final multivariate Cox survival regression model for the duration of cold symptoms – Full Analysis Set | F3 |
| F_14_2_2_2_2_kmcs_fas.rtf | Figure | 14.2.2.2.2 | Kaplan-Meier graph for the duration of cold symptoms by treatment group – Full Analysis Set | F4 |
| T_14_2_2_3_coxqol_fas.rtf | Table | 14.2.2.2.3 | Cox survival regression model for the duration of impact on Quality-of-Life – Full Analysis Set | T15 |
| F_14_2_2_2_3_1_hrqol_fas.rtf | Figure | 14.2.2.2.3.1 | Forest plot of Hazard Ratios from final multivariate Cox survival regression model for the duration of impact on Quality-of-Life – Full Analysis Set | F3 |
| F_14_2_2_2_3_2_kmqol_fas.rtf | Figure | 14.2.2.3.2 | Kaplan-Meier graph for the duration of impact on Quality-of-Life by treatment group – Full Analysis Set | F4 |
| T_14_2_2_3_1_cccmed_fas.rtf | Table | 14.2.2.3.1 | Impact of the treatment on the intake of conventional common cold medications – Full Analysis Set | T16 |
| T 14 2 2 3 2 antibio fas.rtf | Table | 14.2.2.3.2 | Impact of the treatment on the intake of antibiotics – Full Analysis Set | T16 |
| T_14_2_2_3_3_antipyr_fas.rtf | Table | 14.2.2.3.3 | Impact of the treatment on the intake of antipyretics – Full Analysis Set | T16 |
| T_14_2_2_3_4_mucol_fas.rtf | Table | 14.2.2.3.4 | Impact of the treatment on the intake of mucolytics – Full Analysis Set | T16 |
| T 14 2 2 3 5 decong fas.rtf | Table | 14.2.2.3.5 | Impact of the treatment on the intake of decongestants – Full Analysis Set | T16 |
| T_14_2_2_3_6_antitus_fas.rtf | Table | 14.2.2.3.6 | Impact of the treatment on the intake of antitussives – Full Analysis Set | T16 |
| T_14_2_2_3_7_cortico_fas.rtf | Table | 14.2.2.3.7 | Impact of the treatment on the intake of systemic and topical corticosteroids – Full Analysis Set | T16 |
| T_14_2_3_cm_fas.rtf | Table | 14.2.3 | Concomitant treatments – Full Analysis Set | T5 |
| T 14 2 4 1 1 1 ae saf.rtf | Table | 14.2.4.1.1.1 | Summary of non-related adverse events – Safety Set | T17 |
| T 14 2 4 1 1 2 ae fas.rtf | Table | 14.2.4.1.1.2 | Summary of non-related adverse events – Full Analysis Set | T17 |

AXIODIS CRO 28/47

Final version – August 09th, 2023

| File (BASICC) | Type | Number | Title | Mock |
|---|---|---|---|---|
| T_14_2_4_1_2_1_trtae_saf.rtf | Table | 14.2.4.1.2.1 | Non-related treatment-emergent adverse events by System Organ Class and Preferred Term – Safety Set | T18 |
| T_14_2_4_1_2_2_trtae_fas.rtf | Table | 14.2.4.1.2.2 | Non-related treatment-emergent adverse events by System Organ Class and Preferred Term – Full Analysis Set | T18 |
| L_14_2_4_2_1_1_sae_saf.rtf | Listing | 14.2.4.2.1.1 | Serious non-related adverse events – Safety Set | L3 |
| L_14_2_4_2_1_2_sae_fas.rtf | Listing | 14.2.4.2.1.2 | Serious non-related adverse events – Full Analysis Set | L3 |
| L_14_2_4_2_2_1_aedisct_saf.rtf | Listing | 14.2.4.2.2.1 | Non-related adverse events leading to definitive discontinuation of the trial device – Safety Set | L3 |
| L_14_2_4_2_2_2_aedisct_fas.rtf | Listing | 14.2.4.2.2.2 | Non-related adverse events leading to definitive discontinuation of the trial device – Full Analysis Set | L3 |
| L_14_2_4_2_3_1_aediscs_saf.rtf | Listing | 14.2.4.2.3.1 | Non-related adverse events leading to definitive discontinuation of the study – Safety Set | L3 |
| L_14_2_4_2_3_2_aediscs_fas.rtf | Listing | 14.2.4.2.3.2 | Non-related adverse events leading to definitive discontinuation of the study – Full Analysis Set | L3 |
| SAFETY – INCIDENTS | | | | |
| T_14_3_1_1_incsum_saf.rtf | Table | 14.3.1.1 | Summary of incidents – Safety Set | T17 |
| T_14_3_1_2_incsocpt_saf.rtf | Table | 14.3.1.2 | Incidents by System Organ Class and Preferred Term – Safety Set | T18 |
| L_14_3_2_1_sinc_saf.rtf | Listing | 14.3.2.1 | Serious incidents – Safety Set | L3 |
| L_14_3_2_2_incdisct_saf.rtf | Listing | 14.3.2.2 | Incidents leading to definitive discontinuation of the trial device – Safety Set | L3 |
| L_14_3_2_3_incdiscs_saf.rtf | Listing | 14.3.2.3 | Incidents leading to definitive discontinuation of the study – Safety Set | L3 |
| PATIENTS DATA LISTINGS | | | | |
| L_16_2_1_disc.rtf | Listing | 16.2.1 | Discontinued patients | NA |
| L_16_2_2_dv.rtf | Listing | 16.2.2 | Protocol deviations | NA |

AXIODIS CRO 29/47

Study Number: LPH-2202

Statistical Analysis Plan BASICC Final version – August 09th, 2023

| File (BASICC) | Туре | Number | Title | Mock |
|---|---|---|---|---|
| L 16_2_3_excl_eff.rtf | Listing | 16.2.3 | Patients excluded from the efficacy analysis | NA |
| L_16_2_4_1_dm.rtf | Listing | 16.2.4.1 | Demographic characteristics by patient | NA |
| L_16_2_4_2_1_mh.rtf | Listing | 16.2.4.2.1 | Medical history by patient | NA |
| L 16 2 4 2 2 mh coded.rtf | Listing | 16.2.4.2.2 | Medical history events (MedDRA V25.0) | NA |
| L_16_2_4_3_ie.rtf | Listing | 16.2.4.3 | Inclusion/Exclusion criteria | NA |
| L_16_2_4_4_forbidm.rtf | Listing | 16.2.4.4 | Past or concomitant forbidden medications and concomitant treatments for first symptoms of infectious rhinitis at enrolment / inclusion | NA |
| L_16_2_4_5_fever.rtf | Listing | 16.2.4.5 | Fever and body temperature | NA |
| L_16_2_5_1_sv.rtf | Listing | 16.2.5.1 | Dates of visits | NA |
| L_16_2_5_2_rand.rtf | Listing | 16.2.5.2 | Randomization and product unblinding | NA |
| L_16_2_5_3_compl.rtf | Listing | 16.2.5.3 | Compliance to treatment intake | NA |
| L_16_2_6_1_1_arssq.xml | Listing | 16.2.6.1.1 | Acute Rhinitis Symptoms Severity Questionnaire | NA |
| L_16_2_6_1_2_tte.rtf | Listing | 16.2.6.1.2 | Durations of common cold, of cold symptoms and of impacts on Quality-of-Life | NA |
| L_16_2_6_2_1_1 cm.rtf | Listing | 16.2.6.2.1.1 | Previous and concomitant medications by patient | NA |
| L 16 2 6 2 1 2 cm coded.rtf | Listing | 16.2.6.2.1.2 | Coded medications (WHO-DRUG 2022 Q1) | NA |
| L_16_2_6_2_intak.rtf | Listing | 16.2.6.2.2 | Intakes of common cold medications | NA |
| L_16_2_6_2_3_cm_end.rtf | Listing | 16.2.6.2.3 | Concomitant treatments at end of study / premature termination | NA |
| L 16 2 6 3 symp_end.rtf | Listing | 16.2.6.3 | Symptoms of acute rhinitis at end of study / premature termination | NA |
| L_16_2_7_1_ae.rtf | Listing | 16.2.7.1 | Adverse events and incidents | NA |
| L 16 2 7 2 ae coded.rtf | Listing | 16.2.7.2 | Coded adverse events and incidents (MedDRA V25.0) | NA |
| L 16 2 7 3 ae end.rtf | Listing | 16.2.7.3 | Adverse events and incidents at end of study / premature termination | NA |

**AXIODIS CRO** 30/47

# 13.2. Mock tables

# Mock T1

| | Healsea Babykids<br>N=XX | Placebo<br>N=XX | Total<br>N=XX |
|---|---|---|---|
| Analysis Sets | | | |
| Enrolled patients | XX ( XX.X%) | XX ( XX.X%) | XX ( XX.X%) |
| Included patients | XX ( XX.X%) | XX ( XX.X%) | XX ( XX.X%) |
| Randomised patients | XX ( XX.X%) | XX ( XX.X%) | XX (XX.X%) |
| Safety Set | XX ( XX.X%) | XX ( XX.X%) | XX ( XX.X%) |
| Full Analysis Set | XX ( XX.X%) | XX ( XX.X%) | XX (XX.X%) |
| Per Protocol Set | XX ( XX.X%) | XX ( XX.X%) | XX ( XX.X%) |

AXIODIS CRO 31/47

Final version – August 09<sup>th</sup>, 2023

Statistical Analysis Plan

#### Mock F1



AXIODIS CRO 32/47

Study Number: LPH-2202

BASICC

Statistical Analysis Plan
Final version – August 09<sup>th</sup>, 2023

Follow-up: Patients Lost to follow-up (give reasons) (N=XX) {list of patients}

Discontinued intervention (give reasons) (N=XX) {list of patients}

Safety Set (N=XX)

Patients excluded from Safety Set (did not take any treatment) (N=XX) {list of patients}

Full Analysis Set Full Analysis Set (N=XX)

Patients excluded from Full Analysis Set (without any post-baseline efficacy data) (N=XX) {list of patients}

Per Protocol Set Per Protocol Set (N=XX)

Patients excluded from Per Protocol Set (with major protocol deviations) (give reasons) (N=XX) {list of patients}

Healsea Babykids arm

Lost to follow-up (give reasons) (N=XX) {list of patients}

Discontinued intervention (give reasons) (N=XX) {list of patients}

Safety Set (N=XX)

Patients excluded from Safety Set (did not take any treatment) (N=XX) {list of patients}

Full Analysis Set (N=XX)

Patients excluded from Full Analysis Set (without any post-baseline efficacy data) (N=XX) {list of patients}

Per Protocol Set (N=XX)

Patients excluded from Per Protocol Set (with major protocol deviations) (give reasons) (N=XX) {list of patients}

Placebo arm

AXIODIS CRO 33/47

# Final version – August 09<sup>th</sup>, 2023

Statistical Analysis Plan

# Mock T2

| Category of deviation – Type of deviation | Healsea Babykids<br>N=XX | Placebo<br>N=XX | Total<br>N=XX |
|---|---|---|---|
| Patients with at least one protocol deviation | <u> </u> | <u>'</u> | |
| All | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Major deviations | | | |
| All | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| XXXXX | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| XXXXX | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Minor deviations | | | |
| All | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| XXXXX | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| XXXXX | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

# Mock L1

| ID – Sex –<br>Age | Treatment | Safety Set | Full Analysis Set | Per Protocol Set | Protocol deviation | Classification of deviation |
|---|---|---|---|---|---|---|

# Mock T3

| | Healsea Babykids<br>N=XX | Placebo<br>N=XX | Total<br>N=XX |
|---|---|---|---|
| Reason of premature w | ithdrawal | | |
| XXXXXXX | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

# Mock L2

| ID – Sex – Age | Treatment | Safety Set | Full Analysis Set | Per Protocol Set | Reason of withdrawal |
|---|---|---|---|---|---|

AXIODIS CRO 34/47 Study Number: LPH-2202

BASICC

# Mock T4

| | Healsea Babykids<br>N=XX | Placebo<br>N=XX | Total<br>N=XX |
|-------------|--------------------------|-----------------|---------------|
| Age (years) | | | |
| N | XX | XX | XX |
| Missing | XX | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median | XX | XX | XX |
| Q1/Q3 | XX / XX | XX / XX | XX / XX |
| Min/Max | XX / XX | XX / XX | XX / XX |
| Sex | | | |
| N | XX | XX | XX |
| Missing | XX | XX | XX |
| Female | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Male | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

# Mock T5

| ATC1 - ATC2 | Healsea Babykids<br>N=XX | Placebo<br>N=XX | Total<br>N=XX |
|---|---|---|---|
| Patients with at least one previous / concomitant medication | | | |
| All | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| XXXXX | | | |
| All | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| XXXXX | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| XXXXX | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

# Mock T6

| | Healsea Babyki<br>N=XX | ls Placebo<br>N=XX | Total<br>N=XX |
|---|---|---|---|
| Is the patient currently taking antibiotics or has the patie | nt taken antibiotics within 2 weeks before screenin | g? | • |
| N | XX | XX | XX |
| Missing | XX | XX | XX |
| No | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) |
| Yes | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) |
| Is the patient currently taking systemic corticosteroids or | has the patient taken systemic corticosteroids wit | hin 4 weeks before scree | ening? |
| N | XX | XX | XX |
| Missing | XX | XX | XX |
| No | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) |
| Yes | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) |
| Has the patient a chronic use of decongestant? | | | |
| N | XX | XX | XX |
| Missing | XX | XX | XX |
| No | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) |
| Yes | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) |
| Has the patient taken any medicine (in the previous 48 ho | ours) that could modify the ARSSQ assessment? | | |
| N | XX | XX | XX |
| Missing | XX | XX | XX |
| No | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) |
| Yes | XX (XX.X% | ) XX (XX.X%) | XX (XX.X%) |

AXIODIS CRO 35/47

Statistical Analysis Plan Final version – August 09<sup>th</sup>, 2023

# Mock T7

| | Healsea Babykids<br>N=XX | Placebo<br>N=XX | Total<br>N=XX |
|---|---|---|---|
| Has the patient taken / has the patient been prescribed any treatment for first symptoms of | f infectious rhinitis? | | |
| N | XX | XX | XX |
| Missing | XX | XX | XX |
| No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Yes | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

# Mock T8

| SOC - Preferred Term | Healsea Babykids<br>N=XX | Placebo<br>N=XX | Total<br>N=XX |
|---|---|---|---|
| Patients with at least one medical histo | ory | | |
| All | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| XXXXX | | | |
| All | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| XXXXX | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| XXXXX | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

AXIODIS CRO 36/47

Mock T9

| | Healsea Babykids<br>N=XX | Placebo<br>N=XX | Total<br>N=XX |
|---|---|---|---|
| How sick does your child | I feel today? | | |
| N | XX | XX | XX |
| Missing | XX | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median | XX | XX | XX |
| Q1/Q3 | XX / XX | XX / XX | XX / XX |
| Min/Max | XX / XX | XX / XX | XX / XX |
| Between-groups test | XXX (Student/Wilcoxon) | | |
| Runny nose | 1 | <u>'</u> | |
| N | XX | XX | XX |
| Missing | XX | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median | XX | XX | XX |
| Q1/Q3 | XX / XX | XX / XX | XX / XX |
| Min/Max | XX / XX | XX / XX | XX / XX |
| Between-groups test | XXX (Student/Wilcoxon) | | |
| Stuffy nose / Blocked no | 1 | | ı |
| N | XX | XX | XX |
| Missing | XX | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median | XX | XX | XX |
| Q1/Q3 | XX/XX | XX / XX | XX / XX |
| Min/Max | XX / XX | XX / XX | XX / XX |
| Between-groups test | XXX (Student/Wilcoxon) | AATAA | XX/XX |
| Yellow / Green discharg | <u> </u> | | |
| N | XX | XX | XX |
| Missing | XX | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median | XX | XX.X (XX.X)<br>XX | XX |
| Q1/Q3 | XX/XX | XX / XX | XX / XX |
| Min/Max | XX / XX | XX / XX<br>XX / XX | XX / XX |
| | | ΛΛ / ΛΛ | \(\lambda / \lambda \) |
| Between-groups test | XXX (Student/Wilcoxon) | | |
| Nasal crust (dry mucus) | | VV | VV |
| N<br>M: : | XX | XX | XX |
| Missing | XX | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median | XX | XX | XX |
| Q1/Q3 | XX / XX | XX / XX | XX / XX |
| Min/Max | XX / XX | XX / XX | XX / XX |
| Between-groups test | XXX (Student/Wilcoxon) | | |
| Sore throat (hurts to sw | <del>, , </del> | | |
| N | XX | XX | XX |
| Missing | XX | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median | XX | XX | XX |
| Q1/Q3 | XX / XX | XX / XX | XX / XX |
| Min/Max | XX / XX | XX / XX | XX / XX |
| Between-groups test | XXX (Student/Wilcoxon) | | |

AXIODIS CRO 37/47

| | Healsea Babykids<br>N=XX | Placebo<br>N=XX | Total<br>N=XX |
|---|---|---|---|
| Sneezing / Cough | 1 | | ı |
| N | XX | XX | XX |
| Missing | XX | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median | XX | XX | XX |
| Q1/Q3 | XX/XX | XX / XX | XX / XX |
| Min/Max | XX/XX | XX / XX | XX / XX |
| Between-groups test | XXX (Student/Wilcoxon) | | |
| Cold symptoms | , , , | | |
| N | XX | XX | XX |
| Missing | XX | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median | XX | XX | XX |
| Q1/Q3 | XX / XX | XX / XX | XX / XX |
| Min/Max | XX / XX | XX / XX | XX / XX |
| Between-groups test | XXX (Student/Wilcoxon) | AA / AA | AA / AA |
| Impact on Sleeping | AAA (Student Wheoxon) | | |
| N Sleeping | XX | XX | XX |
| N<br>Missing | XX | XX | XX |
| Mean (SD) | | | |
| Median | XX.X (XX.X)<br>XX | XX.X (XX.X)<br>XX | XX.X (XX.X) |
| Q1/Q3 | XX / XX | XX / XX | XX / XX |
| Min/Max | XX / XX | XX / XX | XX / XX |
| Between-groups test | XXX (Student/Wilcoxon) | | |
| Impact on Breathing | | | |
| N | XX | XX | XX |
| Missing | XX | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median | XX | XX | XX |
| Q1/Q3 | XX / XX | XX / XX | XX / XX |
| Min/Max | XX / XX | XX / XX | XX / XX |
| Between-groups test | XXX (Student/Wilcoxon) | | |
| Impact on Playing / Goir | ng to the nursery or to school | | |
| N | XX | XX | XX |
| Missing | XX | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X(XX.X) | XX.X (XX.X) |
| Median | XX | XX | XX |
| Q1/Q3 | XX / XX | XX / XX | XX / XX |
| Min/Max | XX / XX | XX / XX | XX / XX |
| Between-groups test | XXX (Student/Wilcoxon) | | |
| Impact on Quality-of-Li | fe | | |
| N | XX | XX | XX |
| Missing | XX | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| | XX | XX | XX |
| Median | 7121 | | |
| Median<br>Q1/Q3 | XX / XX | XX / XX | XX / XX |
| | | XX / XX<br>XX / XX | XX / XX<br>XX / XX |

AXIODIS CRO 38/47

| | Healsea Babykids<br>N=XX | Placebo<br>N=XX | Total<br>N=XX |
|---|---|---|---|
| N | XX | XX | XX |
| Missing | XX | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median | XX | XX | XX |
| Q1/Q3 | XX / XX | XX / XX | XX / XX |
| Min/Max | XX / XX | XX / XX | XX / XX |
| Between-groups test | XXX (Student/Wilcoxon) | | |

# Mock T10

| | Healsea Babykids<br>N=XX | Placebo<br>N=XX | Total<br>N=XX |
|---|---|---|---|
| Has the patient fever? | | | |
| N | XX | XX | XX |
| Missing | XX | XX | XX |
| No | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Yes | XX (XX.X%) | XX (XX.X%) XX (XX.X%) | |
| Between-groups test | XXX (Chi-2/Fisher) | | |
| Body temperature (°C) | | | |
| N | XX | XX | XX |
| Missing | XX | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median | XX | XX | XX |
| Q1/Q3 | XX / XX | XX / XX | XX / XX |
| Min/Max | XX / XX | XX / XX | XX / XX |
| Between-groups test | XXX (Student/Wilcoxon) | | |

# Mock T11

| | Healsea Babykids<br>N=XX | Placebo<br>N=XX | Total<br>N=XX |
|---|---|---|---|
| Compliance (%) | | | |
| N | XX | XX | XX |
| Missing | XX | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median | XX | XX | XX |
| Q1/Q3 | XX / XX | XX / XX | XX / XX |
| Min/Max | XX / XX | XX / XX | XX / XX |
| Compliance category | | | |
| N | XX | XX | XX |
| Missing | XX | XX | XX |
| <80% | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| [80%; 120%] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| >120% | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

AXIODIS CRO 39/47

# Mock T12

| | Healsea Babykids<br>N=XX | Placebo<br>N=XX | Total<br>N=XX |
|---|---|---|---|
| Study duration (days | ) | | |
| N | XX | XX | XX |
| Missing | XX | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median | XX | XX | XX |
| Q1/Q3 | XX / XX | XX / XX | XX / XX |
| Min/Max | XX / XX | XX / XX | XX / XX |
| Treatment duration ( | days) | | |
| N | XX | XX | XX |
| Missing | XX | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median | XX | XX | XX |
| Q1/Q3 | XX / XX | XX / XX | XX / XX |
| Min/Max | XX / XX | XX / XX | XX / XX |
| Patients who stopped | treatment | · | |
| N | XX | XX | XX |
| Missing | XX | XX | XX |
| Before D8 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| At D8 morning | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| At D8 evening | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| At D9 morning | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| At D9 evening | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| At D10 morning | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| At D10 evening | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| At D11 morning | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| At D11 evening | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| At D12 morning | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| At D12 evening | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| After D12 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

AXIODIS CRO 40/47

Mock T13

| | Healsea Babykids<br>N=XX | Placebo<br>N=XX | Total<br>N=XX |
|---|---|---|---|
| AUC on global score of ARSSQ | | | |
| N | XX | XX | XX |
| Missing | XX | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X(XX.X) | XX.X (XX.X) |
| Median | XX | XX | XX |
| Q1/Q3 | XX / XX | XX / XX | XX / XX |
| Min/Max | XX / XX | XX / XX | XX / XX |
| Between-groups test | XXX (Student/Wilcoxon) | | |

# Mock F2



AXIODIS CRO 41/47

# Mock T14

| | Healsea Babykids<br>N=XX | Placebo<br>N=XX |
|---|---|---|
| AUC on global score of ARSSQ | | |
| ANCOVA model : | | |
| AUC = Treatment + | | |
| Type 3 Tests of Fixed Effects | | |
| Treatment | XXX | |
| | XXX | |
| Adjusted mean | | |
| LSMeans (SE) | XX.X (XX.X) | XX.X (XX.X) |
| [LSM 95%CI] | [XX.X; XX.X] | [XX.X; XX.X] |
| Adjusted mean (diff. vs Placebo) | | |
| LSMeans (SE) | XX.X (XX.X) | |
| [LSM 95%CI] | [XX.X; XX.X] | |
| Contrast vs Placebo, p= | XXX | |

# Mock T15

| | Healsea Babykids<br>N=XX | Placebo<br>N=XX |
|---|---|---|
| Duration of common cold / cold symptoms / impact of | on Quality-of-Life | |
| N | XX | XX |
| Missing | XX | XX |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) |
| Median | XX | XX |
| Q1/Q3 | XX / XX | XX / XX |
| Min/Max | XX / XX | XX / XX |
| Cox survival regression model: | | |
| Hazard Ratios [95%CI] | | |
| Treatment | XX.X [XX.X; XX.X] | |
| | XX.X [XX.X; XX.X] | |
| p-values (Wald) | | |
| Treatment | XXX | |
| | XXX | |

AXIODIS CRO 42/47

Mock F3



For Treatment: the reference is Placebo

AXIODIS CRO 43/47

Mock F4



AXIODIS CRO 44/47

# Mock T16

| | Healsea Babykids<br>N=XX | Placebo |
|----------------------------------|--------------------------|--------------|
| Use of XXX | N=XX | N=XX |
| N | XX | XX |
| Missing | XX | XX |
| No | XX.X (XX.X%) | XX.X (XX.X%) |
| Yes | XX.X (XX.X%) | XX.X (XX.X%) |
| Logistic model : | | , |
| Odds Ratios [95%CI] | | |
| Treatment | XX.X [XX.X; XX.X] | |
| | XX.X [XX.X; XX.X] | |
| p-values (Wald) | | |
| Treatment | XXX | |
| | XXX | |
| Number of days of intakes of XXX | | |
| N | XX | XX |
| Missing | XX | XX |
| 0 | XX.X (XX.X%) | XX.X (XX.X%) |
| 1 | XX.X (XX.X%) | XX.X (XX.X%) |
| 2 | XX.X (XX.X%) | XX.X (XX.X%) |
| | XX.X (XX.X%) | XX.X (XX.X%) |
| Poisson regression : | | |
| Type 3 Tests of Fixed Effects | | |
| Treatment | XXX | |
| | XXX | |

AXIODIS CRO 45/47

# Mock T17

| | Healsea Babykids<br>N=XX | | s Placebo<br>N=XX | | Total<br>N=XX | |
|---|---|---|---|---|---|---|
| | n (%) | [E] | n (%) | [E] | n (%) | [E] |
| Number and percentage of patients with / Number of (non-related) | | | | | | |
| Incident (Adverse event) | XX (XX.X%) | XXX | XX (XX.X%) | XXX | XX (XX.X%) | XXX |
| Incident (Adverse event) leading to definitive study device discontinuation | XX (XX.X%) | XXX | XX (XX.X%) | XXX | XX (XX.X%) | XXX |
| Incident (Adverse event) leading to definitive study discontinuation | XX (XX.X%) | XXX | XX (XX.X%) | XXX | XX (XX.X%) | XXX |
| Serious incident (adverse event) | XX (XX.X%) | XXX | XX (XX.X%) | XXX | XX (XX.X%) | XXX |
| (Treatment-emergent adverse event) | XX (XX.X%) | XXX | XX (XX.X%) | XXX | XX (XX.X%) | XXX |
| (Serious treatment-emergent adverse event) | XX (XX.X%) | XXX | XX (XX.X%) | XXX | XX (XX.X%) | XXX |

# Mock T18

| | Healsea Baby | ykids | Placebo<br>N=XX | | Total<br>N=XX | |
|---|---|---|---|---|---|---|
| SOC - Preferred Term | n (%) | [E] | n (%) | [E] | n (%) | [E] |
| Incidents (Non-related treatment-emergent ad | dverse events) | | | | | |
| All | XX (XX.X%) | XXX | XX (XX.X%) | XXX | XX (XX.X%) | XXX |
| XXXXX | | | | | | |
| All | XX (XX.X%) | XXX | XX (XX.X%) | XXX | XX (XX.X%) | XXX |
| XXXXX | XX (XX.X%) | XXX | XX (XX.X%) | XXX | XX (XX.X%) | XXX |
| XXXXX | XX (XX.X%) | XXX | XX (XX.X%) | XXX | XX (XX.X%) | XXX |

# Mock L3

| ID – Sex – Age | Treatment | Incident (Adverse event) | Start date /<br>end date | Ongoing at the end of the study | Intensity | Serious | Action<br>taken | Causality |
|---|---|---|---|---|---|---|---|---|

AXIODIS CRO 46/47

# 13.3. Acute Rhinitis Symptoms Severity Questionnaire - Daily report

# Q1: How sick does your child feel today: Not sick □ A little sick □ Sick □ Very sick □

# Q2-Q7: How do you evaluate the intensity of the following symptoms of your child?

| Symptoms | Not present | mild | moderate | severe |
|--------------------------------|-------------|------|----------|--------|
| Runny nose | | | | |
| Stuffy nose/blocked nose | 0 | 0 | 0 | 0 |
| Yellow/green<br>discharge | 0 | 0 | 0 | 0 |
| Nasal crust (dry mucus) | 0 | 0 | 0 | 0 |
| Sore throat (hurts to swallow) | 0 | 0 | 0 | 0 |
| Sneezing/cough | | | | |

# Q8-Q10: How do you evaluate the impact of the common cold on your child's activities?

| Activity | No impact | Mild impact | Moderate impact | Severe impact |
|---|---|---|---|---|
| Sleeping | | | | |
| Breathing | | | | |
| Playing/going to the<br>nursery or to school | 0 | 0 | 0 | 0 |

AXIODIS CRO 47/47